CLINICAL TRIAL: NCT03037411
Title: A Real World Evaluation of the ELUVIA Drug Eluting Stent in All-Comers With Superficial Femoral Artery and Proximal Popliteal Artery Disease
Brief Title: A Real World Evaluation of the ELUVIA Stent in Subjects With Lesions Located in the Femoropopliteal Arteries
Acronym: REGAL
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2346
Record Dates: First submitted 2016-12-14; First posted 2017-01-31 (Estimated); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Arterial Occlusive Diseases; Atherosclerosis; Vascular Diseases; Arteriosclerosis
Keywords: Atherosclerosis; Superficial Femoral Artery (SFA); Proximal Popliteal Artery (PPA); Stenting; Paclitaxel; Health Economics
MeSH Terms: conditions — Arterial Occlusive Diseases; Atherosclerosis; Vascular Diseases; Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ELUVIA stent implantation: Peripheral stenting
  Interventions: Device: Peripheral stenting

INTERVENTIONS:
Device: Peripheral stenting — stent implantation during the index procedure

SUMMARY:
The REGAL study is a European, prospective, multi-center Post-Market Clinical Follow-up (PMCF) trial providing additional data including health economics data to support the use of the ELUVIA stent in the treatment of lesions located in the femoropopliteal arteries.

DETAILED DESCRIPTION:
A European, prospective, multi-center Post-Market Clinical Follow-up (PMCF) trial providing additional data including health economics data to support the use of the ELUVIA stent in the treatment of lesions located in the femoropopliteal arteries.

The objective of the study is to collect additional data including health economics data to support the use of the ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and older
2. Subject is willing and able to provide written consent before any study-specific test or procedure is performed and agrees to attend all follow-up visits
3. De novo, restenotic or (re)occluded lesions in the native femoro-popliteal arteries, with reference vessel diameter (RVD) ranging from 4.0-6.0 mm, suitable for endovascular treatment

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant during the course of the study
2. Life expectancy of less than 1 year (which is defined as documented life expectancy less than 12 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the clinical follow-up, limit the subject's compliance with the standard of care follow-up, or impact the scientific integrity of the trial)
3. Known allergy to the ELUVIA stent system or any of its components, concomitant medication, contrast agents (that cannot be medically managed)
4. Subject enrolled in an investigational study that has not reached primary endpoint at the time of enrollment or that clinically interferes with the current study assessments (Note: studies requiring extended follow-up for products that were investigational, but have become commercially available since then are not considered investigational studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Intended population for the REGAL study are 'real world'-patients with symptomatic de-novo, restenotic, or (re)occluded lesions in the native superficial femoral artery (SFA) and/or proximal popliteal artery with reference vessel diameter (RVD) ranging from 4.0-6.0 mm, suitable for endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Health care costs | Index Procedure, 1, 6, 12 and 24 months
  Health care costs at index procedure and changes in health care costs from baseline

SECONDARY OUTCOMES:
Quality of Life Improvement | 1, 6, 12 and 24 months
  Change in EQ-5D-5L™ from baseline
Walking Improvement | 1, 6, 12 and 24 months
  Change in Walking Impairment Questionnaire (WIQ) from baseline
Rate of Primary and Secondary Sustained Clinical Improvement | 1, 6, 12 and 24 months
  Changes in Rutherford Classification from baseline
Rate of Hemodynamic Improvement | 1, 6, 12 and 24 months
  Changes in in Ankle-Brachial Index (ABI) from baseline
Health care utilization | 1, 6, 12 and 24 months
  Changes in healthcare utilization over time

OTHER OUTCOMES:
Technical success of the stenting procedure | During stenting procedure
  Technical success defined as delivery and deployment of the study stent to the target lesion to achieve residual angiographic stenosis no greater than 30% assessed visually
Procedural success of the stenting procedure | within 24 hours of stenting procedure
  Procedural success defined as technical success with no MAEs noted within 24 hours of the stenting procedure
Adverse Event and Major Adverse Event (MAE) rate | 1, 6, 12 and 24 months
  Adverse Event rate and MAE rate, defined as all causes of death, target limb major amputation and/or Target Lesion Revascularization rate at each time point
Primary patency | 6, 12 and 24 months
  Primary patency of target lesion assessed by duplex ultrasound as adjudicated by an independent core laboratory
Clinically-driven Target Lesion Revascularization (TLR) Rate | 1, 6, 12 and 24 months
  Target Lesion Revascularization is defined as any surgical or percutaneous intervention to the target lesion(s) after the stenting procedure
Clinically-driven Target Vessel Revascularization (TVR) Rate | 1, 6, 12 and 24 months
  Target Vessel Revascularization is defined as any surgical or percutaneous intervention to the target vessel after the stenting procedure
Distribution of Rutherford Classification | 1, 6, 12 and 24 months
  Rutherford Classification:
  0 Asymptomatic - Normal Treadmill /stress test
  1. Mild claudication - Completes treadmill exercise; ankle pressure (AP) after exercise <50mm Hg, but >25 mm Hg less than BP
  2. Moderate claudication - Between categories 1 and 3
  3. Severe claudication - Cannot complete treadmill exercise and AP after exercise <50 mm Hg
  4. Ischemic rest pain - Resting AP <40 mm Hg, flat or barely pulsatile ankle or metatarsal pulse volume recording (PVR); toe pressure (TP) <30 mm Hg
  5. Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal edema - Resting AP <60 mm Hg, ankle or metatarsal (MT) PVR flat or barely pulsatile; TP <40 mm Hg
  6. Major tissue loss-extending above MT level - Same as Category 5

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Setacci, Principal Investigator — Policlinico Le Scotte, Siena
Locations (23):
- Medizinische Universität Graz, Graz, Austria
- Belgium (3):
  - ZOL Genk, Genk, Limburg
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen, Vlaams-Brabant
  - CHU Sart Tilman, Liège
- France (2):
  - Centre Hospitalier Universitaire Grenoble-Alpes, Grenoble
  - Clinique Parly II, Le Chesnay
- Italy (7):
  - ASL Asti, Asti
  - Policlinico Vittorio Emanuele, Catania
  - Policlinico di Monza, Monza
  - Policlinico Umberto I, Roma
  - L'Azienda sanitaira ASL Roma 1, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Hospital Azienda Ospedaliera Universitaria Senese, Siena
- Spain (10):
  - Hospital Universitario de Burgos, Burgos
  - Hosp. Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hosp . Universitario de Guadalajara, Guadalajara
  - Hosp. Ntra Sra. del Rosario, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hosp. Complejo Hosp Universitario (CHUO), Ourense
  - Hospital de Montecelo (Pontevedra EOXI), Pontevedra
  - Hospital Parc Tauli, Sabadell
  - Foundation for the Aragonese Healthcare Research Institute, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided